CLINICAL TRIAL: NCT06951724
Title: A Prospective, Multicenter, Randomized Controlled, Noninferiority Clinical Trial Evaluating the Efficacy and Safety of an Aspiration Catheter in Patients Undergoing PCI for Acute ST-Segment Elevation Myocardial Infarction (STEMI)
Brief Title: Coronary Aspiration Catheter Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D23
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Thrombus aspiration therapy using the test device
  Interventions: Device: Aspiration Catheter
- Control Group (Experimental): Thrombus aspiration therapy using the control device
  Interventions: Device: Export Advance Aspiration Catheter

INTERVENTIONS:
Device: Aspiration Catheter — Thrombus aspiration using Aspiration Catheter
  Arms: Test Group
Device: Export Advance Aspiration Catheter — Thrombus aspiration using Export Advance Aspiration Catheter
  Arms: Control Group

SUMMARY:
To evaluation of the efficacy and safety of an aspiration catheter in patients undergoing PCI for acute ST-segment elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

- General inclusion criteria

1. Age 18-80 years old (inclusive);
2. Clinical diagnosis of acute ST-segment elevation myocardial infarction (STEMI) within 24 hours of the onset of the disease (where ST-segment elevation is defined as ST-segment elevation of ≥1mm or 0.1mV in 2 or more consecutive leads of the 12-lead ECG);
3. Voluntary participation and signed written informed consent. Imaging Inclusion Criteria
4. DSA image showed that the target lesion was in situ coronary artery lesion;
5. Target vessel TIMI thrombus load classification ≥ grade 3 and TIMI flow classification ≤ grade 1;

Exclusion Criteria:

- General exclusion criteria

1. previous PCI intervention or coronary artery bypass grafting (CABG) in the target vessel;
2. Comorbid cardiogenic shock;
3. severe renal failure or ongoing dialysis;
4. severe coagulation abnormalities (e.g., hypercoagulability due to blood disorders);
5. Failure of preoperative thrombolysis requiring remedial PCI;
6. Serious bleeding events requiring transfusion therapy within 30 days prior to surgery;
7. Ischemic stroke within 3 months prior to surgery;
8. Known allergy to anticoagulant and antiplatelet agents or contrast media;
9. female subjects who are known to be pregnant or lactating;
10. Participation or planned participation in other clinical studies of drugs or devices;
11. other conditions that the investigator evaluates to be unsuitable for participation in this trial.

    Imaging exclusion criteria
12. Prognostic aspiration catheter needs to pass through the original stent mesh to reach the thrombus aspiration site;
13. severe calcification or tortuosity of the target vessel or extreme angulation that would interfere with the passage of the suction catheter;
14. the presence of an unprotected left main lesion (more than 50% narrowing of the lumen diameter);
15. the presence of severe triple coronary artery lesions requiring revascularization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of TIMI flow grad 3 after PCI | Immediately after procedure
  Defined as the percentage of subjects with TIMI flow graded 3 after PCI.

SECONDARY OUTCOMES:
TIMI flow after PCI | Immediately after procedure
  Target vessel TIMI (Thrombolysis In Myocardial Infarction) flow grad after PCI, after completion of of coronary thrombus using the test device or control device to complete thrombus aspiration
MBG | Immediately after procedure
  MBG (Myocardial Blush Grade) after coronary thrombus aspiration using either the test device or the control device. There are 4 levels of MBG. Grades range from 0 and up to 3, with higher grades being better.
TIMI Thrombus Grade | Immediately after procedure
  TIMI Thrombus Grade after coronary thrombus aspiration using either the test device or the control device. There are 6 levels of MBG. Grades range from 0 and up to 5, with higher grades being worse.
STR(ST-segment resolution) at 90 minutes | Day 0
  The index of change in the highest level of ST-segment elevation relative to the highest level of preoperative ST-segment elevation was assessed on the basis of electrocardiographic at 90 min ± 30 min after PCI.
Thrombus aspiration time and number of aspirations | Immediately after procedure
  Record and compare the total thrombus aspiration time and number of aspirations in both groups.
Device technical success rate | Immediately after procedure
  The test device or control device is able to successfully pass through all target lesions, complete thrombus aspiration, and successfully withdraw without complications relate to the procedure during thrombus aspiration, and TIMI flow grade 3 in the immediately after PCI.
MACE | 30-day follow-up after procedure
  MACE includes cardiovascular death, recurrent myocardial infarction, all strokes, and target vessel revascularization (TVR)
AE and SAE | 30-day follow-up after procedure
  Incidence of all adverse events, serious adverse events in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No